CLINICAL TRIAL: NCT03300440
Title: The Influence of Probiotics on Body and Mind in Individuals With Psychiatric Disorders - a Clinical Study
Brief Title: PROVIT The Influence of Probiotics on Body and Mind in Individuals With Psychiatric Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 29-235 ex 16/17
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Mood Disorders; Depression
MeSH Terms: conditions — Mood Disorders; Depression | interventions — Probiotics; Biotin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Probiotics and vitamin B7
  Interventions: Dietary Supplement: Probiotics and vitamin B7
- Control group (Placebo Comparator): Placebo and vitamin B7
  Interventions: Dietary Supplement: Placebo and vitamin B7

INTERVENTIONS:
Dietary Supplement: Probiotics and vitamin B7 — Powder; Sachet to 3 g (3 g = 1 portion) in lyophilized form (7,5 x 109 CFU) Bacteria strains: Bifidobacterium bifidum W23 Bifidobacterium lactis W51 Bifidobacterium lactis W52 Lactobacillus acidophilus W22 Lactobacillus casei W56 Lactobacillus paracasei W20 Lactobacillus plantarum W62 Lactobacillus salivarius W24 Lactococcus lactis W19 125mg D-Biotin (Vitamin B7) 30 mg of Common horsetail 30 mg of Fish collagen 30 mg of Keratin Matrix: corn starch, maltodextrin, inulin, fructooligosaccharides, plant protein, enzymes
  Other Names: Omnibiotics Stress Repair
  Arms: Intervention group
Dietary Supplement: Placebo and vitamin B7 — Powder; Sachet to 3 g (3 g = 1 portion) in lyophilized form 125mg D-Biotin (Vitamin B7) 30 mg of Common horsetail 30 mg of Fish collagen 30 mg of Keratin Matrix: corn starch, maltodextrin, inulin, fructooligosaccharides, plant protein, enzymes
  Other Names: Biotin
  Arms: Control group

SUMMARY:
The aim of this study is to explore the effects of probiotics in individuals with a clinically relevant depression on psychiatric symptoms and cognition, inflammatory parameters, as well as gene-expression. The study is conducted as a placebo-controlled, randomized, double-blind, prospective, monocentric clinical study, with a two-arm parallel group design. Individuals in the intervention group receive the multispecies probiotics "Omnibiotics Stress Repair" in addition to vitamin B7, while individuals in the control group receive "Placebo" in addition to vitamin B7.

DETAILED DESCRIPTION:
The study takes places at the Medical University of Graz, Department of Psychiatry and Psychotherapeutic Medicine. Individuals that start inpatient treatment at the ward in the first floor of the Department because of a major depressive episode are eligible. After inclusion into the study, the participants are asked to fill in different self-rating questionnaires (Becks-Depression Inventory-II BDI-II, Symptom Checklist-90-Revised SCL-90-R, Manie-Selbstbeurteilungsskala german adaptation of Self-Report manic inventory (SRMI) - MSS, food frequency questionnaire). General data are explored routinely, as well as a diagnostic interview (MINI - mini international neuropsychiatric interview, German version 5.0) is performed during the stay at the hospital. Participants are asked to provide a stool probe as soon as possible.

At the day after admission, fasting blood is taken (100ml). Routine parameters are further analyzed at the local laboratory, while the rest is stored at -80 degree for later analyzes. Afterwards a cognitive test-battery is performed to measure verbal learning and memory, information processing speed, cognitive flexibility and working memory capacity.

After one week a further stool probe is taken, to measure possible changes in dietary habits due to the stay at the hospital. Antidepressive treatment at the hospital is continued as treatment as usual.

At the end participants go through a similar cognitive test battery as at the beginning and are asked to fill in the same self-rating questionnaires. If participants are discharged before day 28 they are given their own preparation and instructed to take it at home in the exact same manner. An outpatient appointment at the end of the preparation intake is arranged to collect the fasting blood and stool sample and to perform the cognitive assessment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mood (affective) disorders (ICD 10 F3xx)
* or neurotic, stress-related and somatoform disorders (ICD 10 F4xx),
* inpatient treatment at the ward in the first floor of the Department of Psychiatry and Psychotherapeutic Medicine in Graz
* written informed consent

Exclusion Criteria:

* acute suicidality and potential dangers for themselves or other persons
* intake of antibiotics during the last month
* intake of food supplement with probiotic cultures or butyrate during the last year
* persons who are incapable of giving consent
* dementia (Mini Mental Status Examination ≤ 20)
* mental retardation
* misuse of laxatives and diuretics
* acute or chronical gastrointestinal infection or diseases
* pregnancy or breastfeeding period
* acute tumor or autoimmune diseases
* organic brain/mental disorders
* active drug or alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-06-21 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Changes in fecal butyrate levels [μmol/g] | 28 (+/- 2) days
  Stool diagnostics is performed by Biovis
Changes in fecal zonulin levels [ng/ml] | 28 (+/- 2) days
  Stool diagnostics is performed by Biovis
Changes in gastrointestinal quality of life [total score] | 28 (+/- 2) days
  Gastrointestinal quality of life index (Eypasch E, Wood-Dauphinée S, Williams JI, et al. The Gastrointestinal Quality of Life Index. A clinical index for measuring patient status in gastroenterologic surgery. Chirurg. 1993;64(4):264-274.)
Changes in depressive symptoms [HAM-D - total score] | 28 (+/- 2) days
  Clinical assessment of Hamilton Rating Scale for Depression (Hamilton, M. A rating scale for depression. Journal of Neurology, Neurosurgery and Psychiatry. 1960;23: 56-62)
Changes in depressive symptoms [BDI-II - total score] | 28 (+/- 2) days
  Self-rating of depressive symptoms by the patient with Beck Depression Inventory-II (Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. Journal of Personality Assessment. 1996;67 (3): 588-97.)
Changes in overall psychological distress [SCL-90-R9 - GSI] | 28 (+/- 2) days
  GSI - global severity index of Symptom Checklist-90-Revised (Franke, GH. SCL-90-R. Die Symptom-Checkliste von Derogatis-Deutsche Version. Göttingen: Beltz, 1995.)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Reininghaus, PD, MD, Principal Investigator — Medical University of Graz, Department of Psychiatry and Psychotherapeutic Medicine
Locations (1):
- Medical University of Graz, Department of Psychiatry and Psychotherapeutic Medicine, Graz, Styria, Austria